CLINICAL TRIAL: NCT01291953
Title: Effectiveness of Early Detection of Atrial Fibrillation in People 65 Years or More bt Physicians and Nurse in Primary Care
Brief Title: Effectiveness of Early Detection of Atrial Fibrillation
Acronym: FAMDAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Collaborators: Spanish Society of Family and Community Medicine (Other)
Responsible Party: Principal Investigator, Luis A Perula, Responsible GIEAP, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PI-0419-2010
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; screening; prevention; case finding; primary care
MeSH Terms: conditions — Atrial Fibrillation | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screening (Experimental): Opportunist Screening asymptomatic patients. Taking the arterial pulse. Will invite patient to realize an ECG, if pulse is irregular
  Interventions: Procedure: Screening
- Control (Active Comparator): Case finding of patient whith symptoms of atrial fibrilation. Taking the arterial pulse. ECG if pulse is irregular
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Screening — Determination of the arterial pulse and if it is arrhythmic, accomplishment of an ECG
  Other Names: Asymptomatic patient
  Arms: Screening
Procedure: Control — Determination of the arterial pulse and if it is arrhythmic, accomplishment of an ECG
  Other Names: Symptomatic patient
  Arms: Control

SUMMARY:
To verify if the screening opportunistic of Atrial Fibrillation (AF) by means of the measurement of the arterial peripheral pulse is more effective than the habitual practice for the early detection of AF in 65-year-old who come to Primary care

ELIGIBILITY:
Inclusion Criteria:

* Patients that come to his center of health for any motive.

  * That give his assent informed to take part in the study.

Exclusion Criteria:

* FA previous Diagnosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6990 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
efficacy of screening: number of cases diagnosed of Atrial fibrillation (AF) | one year
  Risk Relative (RR)=number of cases of AF with the Screening/number of cases of AF with the habitual intervention

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Perula, PhD, Principal Investigator — Andalusian Health Service

REFERENCES:
- [Derived] Gonzalez Blanco V, Perula de Torres LA, Martin Rioboo E, Martinez Adell MA, Parras Rejano JM, Gonzalez Lama J, Ruiz Moruno J, Martin Alvarez R, Fernandez Garcia JA, Ruiz de Castroviejo J, Roldan Villalobos A, Ruiz Moral R; grupo de estudio colaborativo DOFA-AP. Opportunistic screening for atrial fibrillation versus detecting symptomatic patients aged 65 years and older: A cluster-controlled clinical trial. Med Clin (Barc). 2017 Jan 6;148(1):8-15. doi: 10.1016/j.medcli.2016.07.036. Epub 2016 Oct 26. English, Spanish. PMID 28196583
- [Derived] Perula-de-Torres LA, Martinez-Adell MA, Gonzalez-Blanco V, Baena-Diez JM, Martin-Rioboo E, Parras-Rejano JM, Gonzalez-Lama J, Martin-Alvarez R, Ruiz-Moral R, Fernandez-Garcia JA, Perez-Diaz M, Ruiz-de-Castroviejo J, Perula-de-Torres C, Valero-Martin A, Roldan-Villalobos A, Criado-Larumbe M, Burdoy-Joaquin E, Coma-Sole M, Cervera-Leon M, Cuixart-Costa L; Collaborative Group DOFA-AP. Opportunistic detection of atrial fibrillation in subjects aged 65 years or older in primare care: a randomised clinical trial of efficacy. DOFA-AP study protocol. BMC Fam Pract. 2012 Oct 30;13:106. doi: 10.1186/1471-2296-13-106. PMID 23130754
- See also: Study protocol — http://www.biomedcentral.com/1471-2296/13/106